CLINICAL TRIAL: NCT04548492
Title: The Validity of Modern Mobile Applications in Management of COVID-19 Home Isolation Patients: a Randomized Survey for Health Care Professionals
Brief Title: The Validity of Modern Mobile Applications in Management of COVID-19 Home Isolation Patients: a Survey for Health Care Professionals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant professor, Ain Shams University
Other Study IDs: 75 / 2020
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: the Use of Modern Technology Applications in Home Isolation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — to assess and validate how healthcare professionals can trigger or inhibit the use of modern technology applications in home isolation

SUMMARY:
In late 2019, a novel coronavirus, SARS-CoV-2, was identified as the causative agent of a cluster of pneumonia cases (COVID-19) in Wuhan, China. Clinical symptoms of COVID-19 may be mild or severe. The location where a person will self-isolate will be determined by their healthcare provider and their health authority. When determining the location, several factors to determine the suitability of the home setting are described as the case should stay in a room of their own so that they can be isolated from other household members. The rapid increase and evolution of modern mobile applications for communication and messaging for personal purposes have proved great benefit in healthcare management

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals in Ain Shams University, Cairo, Egypt.

Exclusion Criteria:

* junior Staff

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthcare professionals
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
rate of reassurance delivered from doctors to patients through Whatsapp | 3 months